CLINICAL TRIAL: NCT01325987
Title: Vitamin D on Glycemic Control in African American Children With Type 2 Diabetes
Brief Title: African American Children, Glycemic Control, and Type 2 Diabetes
Acronym: ACT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: F101109002
Record Dates: First submitted 2011-03-28; First posted 2011-03-30 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Type 2 Diabetes; Vitamin D Deficiency
Keywords: Type 2 diabetes; Vitamin D deficiency; Glycemic control
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Vitamin D Deficiency | interventions — Ergocalciferols; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- sugar pill (Placebo Comparator): Subjects with vitamin D deficiency (serum 25(OH)D <20ng/ml) will receive an 8 week of vitamin D treatment (50,000 IU oral vitamin D2/once per week) vs. placebo. All subjects will continue their existing hypoglycemic regimen.
  Interventions: Other: Sugar pill
- vitamin D2 (Experimental): Subjects with vitamin D deficiency (serum 25(OH)D <20ng/ml) will receive an 8 week of vitamin D treatment (50,000 IU oral vitamin D2/once per week) vs. placebo. All subjects will continue their existing hypoglycemic regimen.
  Interventions: Dietary Supplement: Vitamin D2

INTERVENTIONS:
Dietary Supplement: Vitamin D2 — Subjects with vitamin D deficiency (serum 25(OH)D <20ng/ml) will receive an 8 week of vitamin D treatment (50,000 IU oral vitamin D2/once per week) vs. placebo. All subjects will continue their existing hypoglycemic regimen.
  Other Names: Group 1: vitamin D2 50000 IU weekly once for 8 weeks
  Arms: vitamin D2
Other: Sugar pill — 1. group: vitamin D2 50000 IU weekly once for 8 weeks
  2. nd group: placebo weekly once for 8 weeks
  Arms: sugar pill

SUMMARY:
Using a randomized, placebo-controlled trial design in subjects with vitamin D deficiency, the investigators propose to determine if vitamin D treatment improves glycemic control in vitamin D deficient subjects with T2DM. The investigators hypothesize that oral vitamin D treatment will improve glycemic control and ß-cell function in vitamin D deficient AA subjects with T2DM. The investigators further hypothesize that maintaining serum 25(OH)D concentrations above 20 ng/ml with oral supplementation of vitamin D will have additional glycemic control effects.

DETAILED DESCRIPTION:
Current literature suggests that 25-hydroxyvitamin D (25(OH)D) is inversely related to risk of type 2 diabetes mellitus (T2DM). African Americans (AA) have significantly less 25(OH)D concentrations, greater chances of poor glycemic control compared to European Americans (EA). The primary objective is to evaluate if the differences in glycemic control in children with type 2 diabetes are explained by differences in serum concentrations of 25(OH)D. A secondary aim is to demonstrate that subjects with vitamin D deficiency (serum 25(OH)D <20ng/ml) and T2DM who receive an 8 week of vitamin D treatment (50,000 IU oral vitamin D2/once per week) have greater improvement than subjects who receive placebo in glycemic control, as measured by HbA1c and endogenous insulin secretion, as assessed by area under the concentration-time curve (AUC) for mixed meal-stimulated C peptide, at 3 months after study drug administration. Research design: Randomized, placebo-controlled, double blind study design in children with T2DM and vitamin D deficiency. Glycemic control will be determined by HbA1C levels, fasting glucose and area under the curve (AUC) for glucose after a mixed meal tolerance test (MMTT). Measures of beta cell function will be determined by AUC for c-peptide and glucose after MMTT. This study is warranted in AA adolescents with T2DM as any positive interventions could have life long impact and will lead to future larger clinical trials.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 DM with acanthosis
* African American
* 12-18 years
* BMI> 85%
* Tanner Stage > 4

Exclusion Criteria:

* Those taking vitamin D
* Pregnancy
* Those with chronic health conditions other than diabetes
* Those who are deemed medically unstable to participate in research

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 31 (Actual)
Dates: Start 2011-03; Primary Completion 2012-12 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
HbA1C | 3 -4 months
  glycemic control

SECONDARY OUTCOMES:
AUC for c-peptide and glucose after MMTT | 3- 4months
  Area under the curve (AUC) for glucose after a mixed meal tolerance test (MMTT)

CONTACTS AND LOCATIONS:
Overall Officials: Ambika Ashraf, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States